CLINICAL TRIAL: NCT07240805
Title: Digital Health Technologies For Monitoring Disease Symptoms in Progressive Supranuclear Palsy and Dementia With Lewy Bodies
Brief Title: Digital Health Technologies for Progressive Supranuclear Palsy and Dementia With Lewy Bodies
Status: Not yet recruiting | Type: Observational
Sponsor: BioSensics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Johns Hopkins University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1UF1AG094587-01 (NIH); 1UF1AG094587-01 (NIH)
Record Dates: First submitted 2025-11-11; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Progressive Supranuclear Palsy(PSP); Dementia With Lewy Bodies (DLB); PSP; Lewy Body Dementia (LBD); Lewy Body Disease
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Lewy Body Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Progressive Supranuclear Palsy (PSP): 30 patients meeting clinical diagnostic criteria for probable Progressive Supranuclear Palsy will be recruited for the study
- Dementia with Lewy Bodies (DLB) and Mild Cognitive Impairment with Lewy Bodies (MCI-LB): 30 patients meeting clinical diagnostic criteria for probable MCI-LB or DLB will be recruited into the study

SUMMARY:
Progressive supranuclear palsy (PSP), mild cognitive impairment with Lewy bodies (MCI-LB), and Dementia with Lewy Bodies (DLB) are severe neurodegenerative diseases that cause significant motor impairment impacting daily function. Researchers at BioSensics, Johns Hopkins School of Medicine, Massachusetts General Hospital and their collaborators aim to conduct an analytical and clinical validation of wearable-based digital health technologies for monitoring upper and lower limb function in PSP, MCI-LB and DLB that could enable frequent, at-home monitoring and be incorporated into future clinical trials.

DETAILED DESCRIPTION:
PSP is a severe and rapidly progressive frontotemporal lobar degeneration (FTLD) syndrome that lacks effective treatment and leads to a rapid onset of dementia, disability, and eventually death. Dementia with Lewy bodies (DLB) is the second most common type of neurodegenerative dementia after Alzheimer's disease that severely impacts daily function and shortens lifespan. Mild cognitive impairment with Lewy bodies (MCI-LB) is an earlier stage where cognitive impairment is noticeable, but does not significantly interfere with living to the degree as seen in DLB. Both PSP and DLB cause significant motor impairment, resulting in progressive loss of independence in activities of daily living, such as eating, dressing, and writing. Despite approximately 200 ongoing clinical trials in PSP and DLB, there are no FDA-approved treatments for FTLD syndromes (including PSP) or DLB. One of the key challenges in the development of new effective therapies for DLB syndromes is the lack of validated instruments and biomarkers to measure disease severity, disease progression, and the effect of therapeutic interventions. Clinical measures of PSP and DLB, largely based on quantitative variations on the neurological exam, have suboptimal sensitivity to change and relevance to clinical meaning in patients' lives. Since 2019, BioSensics, MGH and JHU have partnered to develop a remote monitoring solution for FTLD syndromes using wearable sensors and a series of digital assessments. The solution uses PAMSys, a FDA-listed Class II pendant sensor for monitoring physical activity, posture, and walking parameters during activities of daily living, where the investigators have demonstrated the feasibility of using PAMSys for tracking ambulatory change in PSP. In this project, the investigators will use PAMSys pendant, PAMSys ULM wrist sensors, and PAMSys Gait ankle sensors to enable comprehensive monitoring of upper and lower limb function in PSP and DLB. The will demonstrate the accuracy (analytical validation) of PAMSys, PAMSys ULM and PAMSys Gait sensors in PSP and DLB. Digital speech, fine motor control, and cognitive assessment data will also be collected from the participants using a study tablet. In addition, a proof-of-concept study will be conducted to demonstrate the feasibility and reliability of monitoring motor function in PSP and DLB using the wearable sensors. Clinically, the proposed solution can be used to develop more sensitive approaches to monitor an individual's response to new therapies. Such solutions can enable the detection of subtle changes in movement, ambulation, and motor function while providing specific individualized insights into the clinical phase of disease. Additionally, by testing whether disease outcomes can be measured remotely in patients' homes, this project will be a crucial step forward for both research and clinical care that could meaningfully reduce both financial and time costs for patients, clinicians, researchers, and pharmaceutical companies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 40-89 meeting clinical diagnostic criteria for probable PSP, probable MCI-LB or probable DLB.
* Able to be present for all study procedures, complete questionnaires and assist during home data collection.
* Eligible participants must be fluent in reading and speaking English and must be capable of providing informed consent based on the principal investigator's judgment.
* Must have a caregiver or study partner who is willing and able to assist with all study-related procedures.
* Ambulatory (able to take 10 steps with minimal support such as use of a cane)

Exclusion Criteria:

* Any neurological, medical, or psychiatric condition that would preclude or confound participation in study activities based on the investigator's judgment.
* History of frequent falls defined as more than 5 falls per month, will not be eligible to participate in the study.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with clinical diagnostic criteria for probable PSP, probable MCI-LB or probable DLB
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
2-Minute Walk Test (2MWT) | Baseline.
  Participants will perform the 2-minute walk test (2MWT) while wearing a PAMSys pendant sensor, and two PAMSys Gait ankle sensors.
Timed Up & Go Test (TUG) | Baseline.
  Participants will perform the (TUG) test while wearing a PAMSys pendant sensor, and two PAMSys Gait ankle sensors.
5-times Sit-to-Stand Test (5xSTS) | Baseline.
  Participants will perform the 5-times Sit-to-Stand Test (5xSTS) while wearing a PAMSys pendant sensor.
Box and Block test (BBT) | Baseline.
  Participants will perform the Box and Block test (BBT) while wearing two PAMSys ULM wrist sensors.
9-Hole Peg Test (9HPT) | Baseline
  Participants will perform the 9-Hole Peg Test (9HPT) while wearing two PAMSys ULM wrist sensors.
Physical Activity Monitoring | 14 days
  Following the baseline visit, participants will be asked to wear a PAMSys pendant sensor for 14 days at home. The average daily number of steps will be measured using the PAMSys pendant.
Gait Monitoring | 14 days
  Following the baseline visit, participants will be asked to wear two PAMSys Gait ankle sensors for 14 days at home. Daily average stride velocity will be measured using the PAMSys Gait ankle sensors. The stride velocity unit is m/s.
Hand Function Monitoring | 14 days
  Following the baseline visit, participants will be asked to wear two PAMSys ULM wrist sensors for 14 days at home. Average daily number of hand goal-directed movements will be measured using the AMSys ULM wrist sensors.

SECONDARY OUTCOMES:
Schwab and England Activities of Daily Living (SE-ADL) | Baseline.
  This is a standard patient-reported outcome to measure of functional ability. The SE-ADL scores range from 0%-100%, where 0% represents a worse outcome.
Zaret Burden Interview (ZBI) | Baseline.
  The ZBI is completed by a reliable caregiver. The ZBI scores range from 0-88, where 88 represents a worse outcome.
Symbol Digit Modalities Test (SDMT) | Baseline.
  This brief cognitive test examines processing speed and sustained attention.
Montreal Cognitive Assessment (MoCA) | Baseline.
  This is a brief global cognitive screening assessment. Scores range from 0 to 30 where 0 represents a worse outcome.
Patient Global Impression Scale (PGIS) | Baseline.
  This is a brief patient-reported global assessment of disease severity. Participants rate their condition from 0 (no severity) to 5 (very severe).

OTHER OUTCOMES:
Digital Speech Assessment | Baseline.
  Using a study tablet, participants will perform a series of digital speech assessments. The collected speech data will be analyzed using BioDigit Speech, an automatic speech analysis software developed by BioSensics.
Digital Cognitive Assessment | Baseline.
  Using a study tablet, participants will perform a series of digital cognitive assessments.
Digital Fine Motor Control Assessment | Baseline.
  Using a study tablet, participants will perform a series of tapping tests.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins University School of Medicine, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
All dataset(s) that can be shared will be deposited in NeuroBANK™. NeuroBANK is a patient-centric clinical research platform that allows capture and aggregation of clinical and clinical research data from simultaneously running research projects and links these data with biospecimen repositories, image banks and genetic information. The database is built upon Chapter 21 CFR Part 11 compliant features. NeuroBANK is hosted and maintained by the Center for Innovation & Bioinformatics (CIB) within the Neurological Clinical Research Institute at Massachusetts General Hospital.
Time Frame: Deidentified participant data may be requested after the study has completed data cleaning and analysis, starting in January 2029
Access Criteria: Requests for data from this repository are made through the CIB.

REFERENCES:
- [Background] Nunes AS, Yildiz Potter I, Mishra RK, Bonato P, Vaziri A. A deep learning wearable-based solution for continuous at-home monitoring of upper limb goal-directed movements. Front Neurol. 2024 Jan 5;14:1295132. doi: 10.3389/fneur.2023.1295132. eCollection 2023. PMID 38249724
- [Background] Sharma M, Mishra RK, Hall AJ, Casado J, Cole R, Nunes AS, Barchard G, Vaziri A, Pantelyat A, Wills AM. Remote at-home wearable-based gait assessments in Progressive Supranuclear Palsy compared to Parkinson's Disease. BMC Neurol. 2023 Dec 11;23(1):434. doi: 10.1186/s12883-023-03466-2. PMID 38082255